CLINICAL TRIAL: NCT07002099
Title: Selinexor, High-dose Methotrexate, and Rituximab Combined With Radiotherapy for Newly Diagnosed, Transplant-ineligible Patients With Central Nervous System Lymphoma: An Open-label, Single-arm, Multicenter Phase II Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LK2024097
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Lymphomas
Keywords: Selinexor; central nervous system lymphoma; WBRT
MeSH Terms: conditions — Lymphoma | interventions — selinexor; Methotrexate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Participants in this single-arm study will receive combination therapy as follows:
  Rituximab 375 mg/m² intravenously on Day 0 of each 21-day cycle High-dose Methotrexate (HD-MTX) 3.5 g/m² intravenously over 4 hours on Day 1 of each cycle Selinexor 80 mg orally once weekly (on Days 1, 8, and 15) during each cycle Treatment is administered every 21 days for up to 6 cycles. Tumor response will be evaluated every 3 cycles.
  Patients who achieve a partial response (PR) or better will undergo consolidative low-dose whole-brain radiotherapy (WBRT) at 23.4 Gy in 13 fractions.
  After radiotherapy, patients who maintain a response will continue with maintenance selinexor 80 mg orally once weekly until disease progression, unacceptable toxicity, or withdrawal.
  This arm is designed to assess the synergistic effect of selinexor when combined with standard CNSL chemotherapy and radiotherapy in patients who are not eligible for stem cell transplantation.
  Interventions: Drug: Selinexor + High-dose Methotrexate + Rituximab + WBRT

INTERVENTIONS:
Drug: Selinexor + High-dose Methotrexate + Rituximab + WBRT — Rituximab 375 mg/m² intravenously on Day 0 of each 21-day cycle
  High-dose Methotrexate (HD-MTX) 3.5 g/m² intravenously over 4 hours on Day 1 of each cycle
  Selinexor 80 mg orally once weekly (on Days 1, 8, and 15) during each cycle
  Treatment is administered every 21 days for up to 6 cycles. Tumor response will be evaluated every 3 cycles.
  Patients who achieve a partial response (PR) or better will undergo consolidative low-dose whole-brain radiotherapy (WBRT) at 23.4 Gy in 13 fractions.

SUMMARY:
This phase II clinical trial is designed to evaluate a novel combination treatment for patients with newly diagnosed central nervous system lymphoma (CNSL) who are not candidates for stem cell transplantation. The study will assess the safety and effectiveness of combining selinexor (an oral selective nuclear export inhibitor) with high-dose methotrexate and rituximab chemotherapy, followed by low-dose whole-brain radiotherapy (WBRT). Selinexor has shown promise in enhancing the effects of chemotherapy and radiation in blood cancers.

Patients enrolled in this open-label, single-arm, multicenter study will receive up to six 21-day treatment cycles. Those who respond well will undergo reduced-dose WBRT and continue selinexor as maintenance therapy. The study will measure how many patients respond to the treatment (overall response rate), how long the response lasts (progression-free survival), overall survival, and safety.

This research aims to provide a less toxic and more effective option for treating CNSL in patients who are older or medically unfit for transplantation.

DETAILED DESCRIPTION:
This is a prospective, investigator-initiated, open-label, single-arm, multicenter phase II clinical trial designed to evaluate the efficacy and safety of a combination regimen consisting of selinexor, high-dose methotrexate (HD-MTX), and rituximab, followed by low-dose whole-brain radiotherapy (WBRT), in patients with newly diagnosed primary or secondary central nervous system lymphoma (PCNSL or SCNSL) who are not eligible for autologous stem cell transplantation (ASCT).

Selinexor is a first-in-class, selective inhibitor of nuclear export (SINE) targeting XPO1/CRM1. By blocking nuclear export, selinexor restores nuclear localization and activity of multiple tumor suppressor proteins and growth regulatory factors. Preclinical studies suggest that selinexor may enhance the antitumor activity of chemotherapy and radiotherapy, particularly in hematologic malignancies. Its role in CNSL is supported by its ability to cross the blood-brain barrier and sensitize lymphoma cells to treatment.

Eligible patients will receive six 21-day cycles of combination therapy: rituximab 375 mg/m² IV on day 0, HD-MTX 3.5 g/m² IV over 4 hours on day 1, and selinexor 80 mg orally once weekly (days 1, 8, and 15). Tumor response will be assessed every three cycles. Patients achieving at least partial response (PR) will proceed to consolidative low-dose WBRT (23.4 Gy in 13 fractions), followed by maintenance selinexor (80 mg orally once weekly) until disease progression or unacceptable toxicity.

The primary endpoint is the overall response rate (ORR) based on the Lugano 2014 criteria. Secondary endpoints include complete response rate (CRR), progression-free survival (PFS), overall survival (OS), and safety/tolerability assessed by CTCAE v5.0.

A total of 26 patients will be enrolled. This study aims to provide an effective treatment option for transplant-ineligible CNSL patients and to explore the potential synergistic effects of selinexor with chemotherapy and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female.
2. Histologically confirmed primary CNS lymphoma (PCNSL) or secondary CNS lymphoma (SCNSL) with CNS-only involvement.
3. Ineligible for autologous stem cell transplantation based on clinical assessment or patient refusal.
4. At least one measurable brain lesion ≥1 cm in diameter, or positive cerebrospinal fluid (CSF) cytology/flow cytometry for patients with leptomeningeal disease.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
6. Adequate organ function, including:

   * Absolute neutrophil count (ANC) ≥ 1.0 × 10⁹/L
   * Platelets ≥ 75 × 10⁹/L
   * Hemoglobin ≥ 80 g/L
   * Total bilirubin ≤ 1.5 × ULN (or ≤ 3 × ULN if liver involvement)
   * ALT and AST ≤ 2.5 × ULN (or ≤ 5 × ULN if liver involvement)
   * Creatinine clearance ≥ 30 mL/min (Cockcroft-Gault formula)
   * INR ≤ 1.5 × ULN; APTT within 10 seconds of normal
7. Estimated life expectancy of ≥ 3 months.
8. Negative serum pregnancy test for women of childbearing potential.
9. Ability to understand and willingness to sign a written informed consent form.

Exclusion Criteria:

1. CNS involvement limited to intraocular lymphoma only.
2. Prior systemic therapy for CNS lymphoma.
3. SCNSL with active systemic (non-CNS) disease involvement.
4. Uncontrolled intracranial hypertension.
5. Clinically significant or unstable cardiovascular disease, including:

   * Myocardial infarction within 6 months
   * Unstable angina within 3 months
   * Uncontrolled arrhythmias (e.g., ventricular tachycardia/fibrillation)
   * Congestive heart failure NYHA class ≥ III
   * LVEF < 50% by echocardiography
6. Other severe uncontrolled medical conditions, including active infections requiring systemic therapy.
7. Known active hepatitis B (HBV), hepatitis C (HCV), or HIV infection.
8. Active gastrointestinal dysfunction that interferes with the ability to swallow or absorb oral medication.
9. Prior treatment with selective inhibitor of nuclear export (SINE) compounds, including selinexor.
10. Concurrent malignancy, except for adequately treated basal/squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the cervix, prostate, or breast.
11. Pregnant or breastfeeding women, or subjects unwilling to use medically accepted effective contraception during the study and for 6 months after the last dose.
12. Any condition which, in the investigator's judgment, would make the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  The proportion of participants who achieve a complete response (CR) or partial response (PR) as assessed by investigators according to the 2014 Lugano classification for lymphoma response evaluation.

SECONDARY OUTCOMES:
PFS | 2 years
  Time from enrollment to disease progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Bingzong Li, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Houillier C, Soussain C, Ghesquieres H, Soubeyran P, Chinot O, Taillandier L, Lamy T, Choquet S, Ahle G, Damaj G, Agape P, Molucon-Chabrot C, Amiel A, Delwail V, Fabbro M, Jardin F, Chauchet A, Moles-Moreau MP, Morschhauser F, Casasnovas O, Gressin R, Fornecker LM, Abraham J, Marolleau JP, Tempescul A, Campello C, Colin P, Tamburini J, Laribi K, Serrier C, Haioun C, Chebrek S, Schmitt A, Blonski M, Houot R, Boyle E, Bay JO, Oberic L, Tabouret E, Waultier A, Martin-Duverneuil N, Touitou V, Cassoux N, Kas A, Mokhtari K, Charlotte F, Alentorn A, Feuvret L, Le Garff-Tavernier M, Costopoulos M, Mathon B, Peyre M, Delgadillo D, Douzane H, Genet D, Aidaoui B, Hoang-Xuan K, Gyan E. Management and outcome of primary CNS lymphoma in the modern era: An LOC network study. Neurology. 2020 Mar 10;94(10):e1027-e1039. doi: 10.1212/WNL.0000000000008900. Epub 2020 Jan 6. PMID 31907289
- [Background] Walker JS, Garzon R, Lapalombella R. Selinexor for advanced hematologic malignancies. Leuk Lymphoma. 2020 Oct;61(10):2335-2350. doi: 10.1080/10428194.2020.1775210. Epub 2020 Jun 14. PMID 32536290
- [Background] Neupane K, Wahab A, Masood A, Faraz T, Bahram S, Ehsan H, Hannan A, Anwer F. Profile and Management of Toxicity of Selinexor and Belantamab Mafodotin for the Treatment of Triple Class Refractory Multiple Myeloma. J Blood Med. 2021 Jul 1;12:529-550. doi: 10.2147/JBM.S317966. eCollection 2021. PMID 34234609
- [Background] Lurain K, Uldrick TS, Ramaswami R, Polizzotto MN, Goncalves PH, Widell A, Steinberg SM, Jaffe ES, Pittaluga S, Wang HW, Yuan CM, Tamula MA, Martin S, Wolters PL, George J, Little RF, Yarchoan R. Treatment of HIV-associated primary CNS lymphoma with antiretroviral therapy, rituximab, and high-dose methotrexate. Blood. 2020 Nov 5;136(19):2229-2232. doi: 10.1182/blood.2020006048. No abstract available. PMID 32609814
- [Background] Gandhi MK, Hoang T, Law SC, Brosda S, O'Rourke K, Tobin JWD, Vari F, Murigneux V, Fink L, Gunawardana J, Gould C, Oey H, Bednarska K, Delecluse S, Trappe RU, Merida de Long L, Sabdia MB, Bhagat G, Hapgood G, Blyth E, Clancy L, Wight J, Hawkes E, Rimsza LM, Maguire A, Bojarczuk K, Chapuy B, Keane C. EBV-associated primary CNS lymphoma occurring after immunosuppression is a distinct immunobiological entity. Blood. 2021 Mar 18;137(11):1468-1477. doi: 10.1182/blood.2020008520. PMID 33202420
- [Background] Ostrom QT, Cioffi G, Waite K, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2014-2018. Neuro Oncol. 2021 Oct 5;23(12 Suppl 2):iii1-iii105. doi: 10.1093/neuonc/noab200. PMID 34608945